CLINICAL TRIAL: NCT03771274
Title: Visual Outcomes of an Extended Depth of Focus (EDOF) Intraocular Lens (IOL) Combined With a Multifocal (MF) IOL
Brief Title: Tecnis ZLB00 & Symfony Intraocular Lens Combination Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other); Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP18-002
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Cataract Bilateral; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Tecnis ZLB00 & Symfony IOL (Experimental): The Tecnis multifocal ZLB00 and the Symfony IOLs are presbyopia correcting lenses designed to improve the vision at distance, intermediate and near reducing the need for glasses in patients undergoing cataract surgery.
  Interventions: Device: Tecnis ZLB00 & Symfony IOL

INTERVENTIONS:
Device: Tecnis ZLB00 & Symfony IOL — The Symfony IOL will be implanted in the dominant eye while the Tecnis ZLB00 will be implanted in the non-dominant eye.

SUMMARY:
Current visual outcomes expectations of cataract patients are similar to those of refractive surgery patients. Their desire is to be spectacle independent for far, intermediate and near vision activities. Some may have already enjoyed freedom from glasses and would like to continue after the cataracts are removed. Different options are available. These options include: mono-vision and presbyopia correcting intraocular lenses (IOL). Presbyopia correcting IOLs include accommodative, multifocals and extended depth of focus (EDOF) IOLs. In a previous study, the visual outcomes of the EDOF Toric IOL were evaluated when both eyes were targeted for plano and when the non-dominant eye was set for a small residual myopic error (-0.50 D) or nanovision in patients with astigmatism. The nanovision approach, appeared to provide similar binocular acuity at distance and intermediate but better acuity at near. The purpose of this study is to evaluate the visual outcomes of an EDOF IOL when combined with a multifocal IOL with a +3.25 D add in patients with or without astigmatism undergoing routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing bilateral cataract extraction with intraocular lens implantation.
2. Willing and able to provide written informed consent for participation in the study
3. Willing and able to comply with scheduled visits and other study procedures.
4. Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6-15 days between surgeries.
5. Subjects who require an IOL power in the range of +5.0 D to +34.0 D only.
6. Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

1. Contraindication for a presbyopia correcting IOL.
2. Subjects with severe astigmatism in the non-dominant eye
3. Uncontrolled diabetes.
4. Use of any systemic or topical drug known to interfere with visual performance.
5. Contact lens use during the active treatment portion of the trial.
6. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
7. Clinically significant corneal dystrophy
8. History of chronic intraocular inflammation.
9. History of retinal detachment.
10. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
11. Previous intraocular surgery.
12. Previous refractive surgery.
13. Previous keratoplasty
14. Severe dry eye
15. Pupil abnormalities
16. Subject who may reasonably be expected to require a secondary surgical intervention at any time during the study (other than yttrium aluminum garnet (YAG) capsulotomy, i.e. LASIK)
17. Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
18. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
19. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tecnis ZLB00 & Symfony IOL
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tecnis ZLB00 & Symfony IOL
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Binocular Uncorrected Near (40 cm) Visual Acuity.
Description: Visual acuity measured at 40 cm without wearing any correction.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Tecnis ZLB00 & Symfony IOL
Number analyzed (Participants) | 39
logMAR | 0.13 (0.09)

2. Secondary Outcome: Patient Visual Satisfaction After Cataract Surgery: Questionnaire
Description: Patient's overall satisfaction with their vision after cataract surgery assessed by asking the following question: "Taking all things into account, how satisfied or dissatisfied are you with your vision WITHOUT glasses or contacts with your near vision". Possible answers are: Completely satisfied and mostly satisfied, moderately satisfied, a little satisfied or not at all satisfied.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tecnis ZLB00 & Symfony IOL
Number analyzed (Participants) | 39
Participants
  Completely or mostly satisfied | 27
  Moderately satisfied | 5
  A little or not satisfied | 7

3. Secondary Outcome: Spectacle Independence: Questionnaire
Description: Patient's spectacle independence was assessed using the "Patient Reported Spectacle Independence Questionnaire (PRSIQ) which includes the following questions: 1. During the LAST 7 DAYS, did you need glasses or contacts for near. Possible answers: Yes No.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tecnis ZLB00 & Symfony IOL
Number analyzed (Participants) | 39
Participants
  Yes | 12
  No | 27

4. Secondary Outcome: Number of Participants With Visual Symptoms
Description: Number of participants who reported any visual disturbances or symptoms. One participant could report more than one symptom.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tecnis ZLB00 & Symfony IOL
Number analyzed (Participants) | 39
Participants
  Halos : Yes | 25
  Halos : No | 14
  Sensitivity to light: Yes | 23
  Sensitivity to light: No | 16

ADVERSE EVENTS:
Time Frame: 3 to 5 months
Description: Adverse events were collected from the moment participant signed the informed consent until he or she exited the study.
Arm/Group | Tecnis ZLB00 & Symfony IOL
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT03771274/Prot_SAP_000.pdf